CLINICAL TRIAL: NCT06643676
Title: Effect of Targeted Endodontic Microsurgery on Quality of Life and Healing on Mandibular Molars : A Randomized Controlled Trial
Brief Title: Effect of Targeted Endodontic Microsurgery on Quality of Life and Healing on Mandibular Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Muzaffar Khan
Record Dates: First submitted 2024-07-12; First posted 2024-10-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Periapical Diseases; Periapical Periodontitis; Periapical Cyst; Periapical Granuloma; Periapical Pathology; Endodontic Microsurgery; Targeted Endodontic Microsurgery
MeSH Terms: conditions — Periapical Diseases; Periapical Periodontitis; Radicular Cyst; Periapical Granuloma | interventions — Apicoectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Endodontic Microsurgery using trephine drill and 3d printed surgical guide (Experimental): Endodontic Microsurgery using 3d printed static surgical guide using patient's cbct data
  Interventions: Procedure: Targeted Endodontic Microsurgery Using 3d Printed surgical guide using the patient's CBCT data
- Conventional Endodontic microsurgery using burs (Active Comparator): Conventional Endodontic microsurgery using carbide bur and free hand conventional procedure
  Interventions: Procedure: Conventional Endodontic Microsurgery with a free hand procedure using bur and CBCT analysis

INTERVENTIONS:
Procedure: Targeted Endodontic Microsurgery Using 3d Printed surgical guide using the patient's CBCT data — Patients with apical periodontitis with intact cortex in madibular molars receiving Targeted Endodontic surgery or Guided Endodontic Microsurgery with surgical guide fabricated using the cbct data following failure of non surgical root canal treatment
  Other Names: periapical surgery, Targeted Endodontic Microsurgery, Guided Endodontic Microsurgery; apicoectomy
  Arms: Targeted Endodontic Microsurgery using trephine drill and 3d printed surgical guide
Procedure: Conventional Endodontic Microsurgery with a free hand procedure using bur and CBCT analysis — A conventional endodontic microsurgery using arbitrary localisation technique using the cbct data and performing the surgery with a carbide bur.
  Arms: Conventional Endodontic microsurgery using burs

SUMMARY:
Targeted endodontic microsurgery represents precise and advanced approach to resolving persisting chronic periapical periodontitis after non- surgical root canal treatment. This specialised procedure involves accessing the root tip of the tooth under high magnification using dental operating microscopes and employing microsurgical instruments to remove infected or inflamed tissue, as well as any pathological lesions present in the periapical region. Targeted Endodontic Microsurgery is useful for osteotomy and root- end resection when exacting control of depth, diameter, and angulation of osteotomy and root end resection is necessary. Using a CBCT(cone beam computed tomography) designed 3D - printed surgical guideis a more accurate method for access to the apical portion of the root during surgical endodontics compared with a "freehand" CBCT - approximated conventional method. These guided have the potential to increase accuracy and precision and to reduce intraoperative time as well as postoperative complications. Additionally, it provides a viable treatment option for patients who may not be candidates for traditional root canal therapy or retreatment due to anatomical complexities or previous treatment failures.

DETAILED DESCRIPTION:
Conventional Endodontic microsurgery takes use of a preoperative scan and manual drilling of the osteotomy site with arbitrary measurements followed by retropreparation and forming the apical seal. One of the most critical disadvantages of conventional root-end resection include the damage to anatomically vital structures such as inferior dental nerve, mental nerve, adjacent root and maxillary sinus. In contrast, endodontic microsurgery using the guide template significantly reduces these damages. Pinsky et al confirmed in their in vitro study that the greater accuracyand consistency was achieved during endodontic surgery with surgical guidance without damaging vital structures. An error greater than 3 mm occurred over 22% of the time with freehand whereas none of errors occurred with surgical guidance.

Consequently, targeted endodontic microsurgery has garnered increasing attention as a viable alternative, offering a refined and precise approach to address such challenges.

Even the most skilled surgeons may find endodontic microsurgery difficult. Some medical professionals steer clear using freehand (FH) Endodontic microsurgery in regions where there is a chance of harming important anatomical features including the maxillary sinus, the mental foramen, and arteries. It is Perceived as complex sites include those with limited access, no direct sight, and areas where the apex is placed distant from the buccal cortical bone without any cortical plate fenestratio. Surgeons may be able to perform precise procedures in difficult-to-reach regions with guided Endodontic Microsurgery

Guided Endodontic Microsurgery is virtually planned on 3D software on the preoperative CBCT scan, and the surgeon executes the osteotomy and root-end resection (RER) under static or dynamic navigation.

Static navigation requires a customized 3D-printed surgical guide (3D-SG) to guide the drilling duringosteotomy and RER. Surgical guides contain a guide template that refers to the 3D location of the virtual Endodontic Microsurgery planned in the CBCT to drill accurately Prior research has demonstrated that 3D-SG can reduce the risk of intra-operative complications whileincreasing the precision and effectiveness of EMS. In comparison to free hand Endodontic Microsurgery, guided Endodontic Microsurgery with 3D-Surgical Guide shortens the surgical time, provides superior control over the resection level and bevel off the root, and enables a tailored osteotomy size.

Trephine burs have been used for the removal of failed implants and autogenous bone graft harvesting but have not previously been described in Endodontic Microsurgery .

Targeted Endodontic Microsurgery produces a single-step osteotomy; root-end resection; and biopsy with a defined perforation site, angulation, depth, and diameter. Previous reports have used 3D Surgical Guides to locate an ideal bone perforation site, but none have used trephine burs within a stent to define all parameters of osteotomy and root-end resection.

Also, no clinical study assessing the targeted approach of endodontic microsurgery with Oral health related quality of life has been done. Some of the RCT's are conducted assessing quality of life in patients after conventional periapical surgery, only two retrospective studies considering .Targeted Endodontic Microsurgery have been done and a lack of RCTs comparing targeted Endodontic Microsurgery with conventionalEMS warrants further research.

The aim of this study is to compare the effect of a static computer-aided surgical technique using a 3D- printed guide with a fully guided drill protocol on Oral Health Related Quality of Life against the conventional endodontic microsurgery in mandibular molars.

ELIGIBILITY:
Inclusion Criteria:

* Patients in which non-surgical retreatment is unfeasible (post, anatomical complexity, iatrogenic errors) or previously failed treatment.
* Patients with persistent symptomatic apical periodontitis and periapical radiolucency.
* Tooth with a peri-radicular lesion of strictly endodontic origin (chronic apical periodontitis) and combined endodontic periodontic lesions with the size of lesion ≥5mm.

Patients between 18-55 years of age.

* No general medical contraindications for oral surgical procedures (ASA-1 and ASA-2 according to the classification of the American Society of Anesthesiologists)
* ASA 1- A normal healthy patient. Example: Fit, nonobese (BMI under 30), nonsmoking patient with good exercise tolerance.
* Tooth with adequate final restoration without clinical evidence of coronal leakage.
* No spontaneous pain or swelling.
* Good periodontal health condition at tooth level
* Able to completely understand and sign an informed consent form

Exclusion Criteria:

* Patients with systemic diseases (diabetes mellitus, uncontrolled hypertension grade III, hepatic/renal disease, or systemic bleeding disorders)
* Patients on anticoagulant/ antiplatelet drugs.
* Fractured/perforated teeth.
* Teeth with deep pockets (probing depth > 4 mm).
* Presence of vertical root fracture.
* Miller class III/IV mobility.
* Pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life following periapical surgery | 1 year
  Quality of life quantified using Questionnaire to both groups

SECONDARY OUTCOMES:
Radiographic healing | 1 year
  two dimensional radiographic healing by rud and molten criteria three dimensional radiographic healing with Cbct by modified Penn criteria
Time Taken for surgery | one year
  Time taken to complete surgery in both the groups
Accuracy of surgical access | one year
  Assessment of surgical access accuracy using CBCT-based root length measurement Surgical access accuracy was assessed by comparing preoperative and postoperative root length measurements obtained from cone-beam computed tomography (CBCT) scans in both the targeted endodontic microsurgery (TEMS) and conventional endodontic microsurgery (CEMS) groups. Preoperative CBCT scans were acquired using a limited field of view with standardized imaging parameters and exported in DICOM format for analysis.
  The DICOM datasets were imported into Mimics software (Materialise, Leuven, Belgium) for three-dimensional reconstruction. The involved mandibular molar and the corresponding root were segmented using thresholding and region-growing tools. The long axis of the root was established by connecting the center of the root canal in the coronal third to the anatomical root apex. Preoperative root length was measured as the linear distance from the most apical point of the root apex to a standardized c

CONTACTS AND LOCATIONS:
Overall Officials: Jigyasa grover, MDS, Study Director — PGIDS ROHTAK, HARYANA; sanjay Tewari, MDS, Study Chair — PGIDS ROHTAK HARYANA; MOHAMMED MUZAFFAR KHAN, BDS, Principal Investigator — PGIDS ROHTAK HARYANA
Locations (1):
- Post Graduate Institute of Dental Sciences , Rohtak, Rohtak, Haryana, India